CLINICAL TRIAL: NCT02522260
Title: OptiTrain - Optimal Training for Women With Breast Cancer During Chemotherapy Treatment
Brief Title: OptiTrain - Optimal Training Women With Breast Cancer
Acronym: OptiTrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Yvonne Wengstrom, OCN, PhD, Professor of Nursing, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YWengstrom
Record Dates: First submitted 2015-06-09; First posted 2015-08-13 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Well Being
Keywords: Breast cancer, chemotherapy, symptoms, optimal training
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Active Comparator): Intervention Strength/aerobic exercise, weights, bike or treadmill
  Interventions: Other: Resistance and aerobic training
- Group 2 (Active Comparator): Intervention Aerobic exercise, bike or treadmill
  Interventions: Other: Aerobic training
- Group 3 (Active Comparator): Standard supportive care
  Interventions: Other: Standard supportive care

INTERVENTIONS:
Other: Resistance and aerobic training — Group 1) includes strength exercise of the large muscle groups (2-3 sets, 8-12 repetitions on an intensity of 80 % of 1-RM) and 3x3 min high intensity aerobic exercise (16-18 on Borg scale) on an exercise bike or treadmill twice a week for 16 weeks
  Arms: Group 1
Other: Aerobic training — Group 2) includes aerobic exercise on an exercise bike or treadmill, 20 min moderate intensity (13-15 on Borg scale), and 3x3 min high intensity (16-18 on Borg scale) twice a week during 16 weeks
  Arms: Group 2
Other: Standard supportive care — Standard supportive care
  Arms: Group 3

SUMMARY:
This study on women with breast cancer during and after chemo- and hormonal therapy compares the effect of different physical training programs on physical and mental well-being and systemic inflammation mechanisms in blood. In a sub-group of participants, mitochondrial biogenesis and function and other molecular processes in skeletal muscle biopsies are studied. The women will be randomly allocated into three different intervention arms, a control arm with usual care and two different training arms. All participants will respond to questionnaires and have blood samples and taken and for a subgroup muscle biopsies before and after the exercise intervention. Participants will be supported to uphold exercise through collaboration with Friskis & Svettis and followed for 5 years. Some of the women will also be asked to participate in an in depth interview about the experiences of exercise during ongoing treatment. This study will contribute to increased knowledge about the type, intensity and frequency of training that patients with breast cancer benefit most from with regards to impact on physical and mental wellbeing. This knowledge is of great importance since experience shows that patients and relatives often seek information about rehabilitation, self-care and physical activity. The study will also contribute to the improvement of the patients´ quality of life, ability to return to work, and reduce social costs, but above all, increase the possibility for development and implementation of evidence-based rehabilitation of women with breast cancer during and after active treatment.

DETAILED DESCRIPTION:
Purpose The main aim is to, in women undergoing chemotherapy for breast cancer, explore how different training interventions impact physical capacity and psychological well being.

Research questions

* Does PA improve the ability to return to work after breast cancer treatment is completed?
* How do women with breast cancer during chemotherapy treatment respond to controlled and supervised aerobic fitness training and a combination of aerobic fitness training and strength training in physiological, structural and molecular outcome measures such as muscular strength, aerobic fitness, muscle mass, mitochondrial density, gene activity in muscle and B-Hb, s-CRP and other blood variables,?
* Is there a difference between the women in the aerobic exercise training group, the combined aerobic and strength-training group and the control group regarding symptom distress and health related quality of life?
* Are there any effects of exercise training on chemotherapy completion and hospitalization rates?
* Is adherence to physical exercise impacted by the individuals' personality?
* Are there any remaining effects of the physical exercise intervention, on cardiotoxicity, cognitive function, survival and morbidity, up to 5 years after treatment is completed?
* Is the intervention cost-effective?

Study design and methods Participants A total of 240 women will be recruited from the Department of Oncology Breast and Sarcoma units at Radiumhemmet and Södersjukhuset, Karolinska University Hospital.

Inclusion criteria: patients up to 70 years with breast cancer Stage I-IIIa before the start of chemotherapy. Exclusion criteria: patients with advanced disease, patients where physical activity is considered contraindicated because of medical reasons such as heart or lung disease, brain or bone metastases, cognitive dysfunction, and patients who do not speak or understand the Swedish language.

Randomization The Clinical Trials Unit (KPE) at Radiumhemmet, Karolinska Universitetssjukhuset, conducts inclusion to the study and randomization. The participants are allocated to either two different training groups or a control group. The participants are also randomized to a muscle biopsy (n=45) before and after the intervention.

Group 1) includes strength training of the large muscle groups (2-3 sets, 8-12 repetitions on an intensity of 80 % of 1-RM) and 3x3 min high intensity aerobic exercise (16-18 on Borg scale) on an exercise bike or treadmill twice a week for 16 weeks.

Group 2) includes aerobic exercise on an exercise bike or treadmill, 20 min of moderate intensity (13-15 on Borg scale), and 3x3 min high intensity aerobic exercise (16-18 on Borg scale) twice a week during 16 weeks.

Group 3) control group, will get standard information around physical activity during treatment but no supervised training.

Data Collection Data will be collected for all study participants regarding demographics and diagnosis, cancer treatment, laboratory and sick leave data (patient-reported), relapse, survival, co-morbidity and cause of death in relevant registers.

* Data collection of demographic data occurs before (before randomization) and after the intervention, and at three time points: 1 year, 2 years and 5 years after treatment is completed. Baseline is about 5 weeks after surgery and before initiation of chemotherapy.
* All participants that accept participation in the study will undergo a resting ECG examination and will provide responses to a small, targeted set of heart disease history questions.
* Muscular strength is measured with the instrument JAMAR that is a dynamometer, measuring muscle strength in the hand. Lower limb muscle strength is measured through isometric mid-thigh pull. This is assessed in all study participants at all time points: before and the intervention, year 1, 2, and 5.. The instruments have good reliability and validity.
* Before and after the intervention aerobic fitness (VO2-max) of the participants in the intervention groups will be assessed with a submaximal exercise test. This will be measured at all time points: before and the intervention, year 1, 2, and 5.
* Algometry, to measure pain sensitivity will be performed at time points: before and after the intervention, year 2 and 5.
* Chemotherapy completion, hospitalization, hemoglobin-, lymphocyte- and platelet concentrations during chemotherapy will be extracted from the patients' medical records.
* Blood sampling and muscle biopsy procedures will take place at the KPE lab Radiumhemmet, Karolinska University Hospital, Solna. Muscle biopsies will be obtained under local anesthesia in the m. vastus lateralis (approximately 100 mg) with a Bergström needle. This takes place before the intervention starts and 48-72 hours after the last training session. Mitochondrial density and muscle morphology will be analyzed. Venous blood is sampled at time points: before and the intervention, year 1, and 5, for analysis of white cell distribution, for markers of systemic inflammation, and markers of cardiac damage
* Physical activity level and energy consumption is determined by ActiGraph GT3X (Actigraph). Actigraph is a combined heart rate sensor and accelerometer that continuously collects data. The method has been previously tested and is shown to have good reliability and validity. In this project all the participants in the three groups will be carrying an Actigraph for seven days, before the intervention. An Activity Diary for daily subjective reporting of physical activity will also be used during the intervention period.

Instruments

* Piper Fatigue Scale assesses fatigue in four dimensions. The scale has been shown to have psychometric properties that are reliable for assessing subjective dimensions of fatigue among Swedish populations of cancer patients. Data will be collected for all study participants (intervention and control) before randomization and after the intervention, and at 1 year, 2 years and 5 years after treatment.
* Memorial Symptom Assessment Scale (MSAS) assesses 32 common cancer-related symptoms. The instrument is validated for Swedish patients with breast cancer. Data will be collected for all study participants before randomization and after the intervention, and at 1 year, 2 years and 5 years after treatment.
* EORTC QLQ-C30 is a cancer-specific instrument that measures health-related quality of life in terms of physical, emotional, social, cognitive and everyday function. Data will be collected for all study participants before randomization and after the intervention, and at 1 year, 2 years and 5 years after treatment.
* Sense of coherence (SOC) is a questionnaire, which shows how a person sees the world and his own life as comprehensible, manageable and meaningful. Individuals with a strong sense of coherence are able to mobilize the resources to manage their health during illness and treatment. SOC short version consists of l3 questions that all participants complete once before the start of treatment. The Swedish version of the SOC-13 has been shown to have good validity and reliability. It has also demonstrated high internal consistency.
* The Amsterdam Cognition Scan- an online neuropsychological test battery that measures a broad variety of cognitive functions, measured five years following inclusion to the exercise intervention
* Echocardiogram- to measure cardiac function, five years following inclusion to the exercise intervention

Qualitative interviews

• Individual interviews about/around the experience of physical activity associated with chemotherapy treatment will be carried out with 15 participants. An open question will be asked, such as "Can you describe how you experienced the period of training?". Because of the nature of this question, the women will have the freedom to narrate their stories, and the interview will focus on elements that surface as significant. Supplementary questions will be asked to create depth and further understanding of the phenomena.

Data Analysis Muscle and blood analysis: From 45 participants in the project, we plan to take a muscle biopsy before and after the training intervention. The molecular exercise physiology lab is fully equipped to store muscle biopsies and other biological material. Many methods are set-up in our muscle lab and others are performed in different core facilities. Molecular and biochemical analyses: Skeletal muscle biopsy samples are obtained with the percutaneous needle technique. Analysis of protein content, CS activity, and immunohistochemistry will be performed.

Quantitative Collected quantitative data will be analysed using parametric statistics for normally distributed data and non-parametric statistics for non-normally distributed data. Subgroup analysis will be conducted with a focus on the type of treatment. Power Calculation: variable cancer related fatigue, selected significance level 0.05, power 0.80 = 240 patients will be recruited in total to detect a statistical difference with medium effect size.

Qualitative Qualitative data from individual interviews with 15 patients will be analyzed inductive with content analysis.

Workplan Data collection is currently ongoing and 80 patients are included in the study. With the current inclusion rate the 240 participants will be included by the end of 2015.

To support the women to uphold PA after treatment is completed a collaboration has been initiated with Friskis & Svettis in Stockholm, during the five year follow up period this will encompass FaR (physical activitiy receipt) and invitations to motivational healthy life style sessions three times a year, the sessions will also include information on longterm effects/symptoms of treatment and support with self care.

ELIGIBILITY:
Inclusion Criteria:

patients up to 70 years with breast cancer Stage I-IIIa before the start of chemotherapy.

Exclusion Criteria:

patients with advanced disease, patients where physical activity is considered contraindicated because of medical reasons such as heart or lung disease, brain or bone metastases, cognitive dysfunction, and patients who do not speak or understand the Swedish language.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Cancer related fatigue | Change from baseline to 16 weeks, 1 year, 2 years, and 5 years post baseline
  Piper fatigue scale

SECONDARY OUTCOMES:
Health Related Quality of Life | Change from baseline to 16 weeks, 1 year, 2 years, and 5 years post baseline
  EORTC-QLQ-C30
Symptoms | Change from baseline to 16 weeks, 1 year, 2 years, and 5 years post baseline
  Memorial Symptom Assessment Scale
Pain sensitivity | Change from baseline to 16 weeks, 2 years and 5 years post baseline
  Algometer
Aerobic fitness | Change from baseline to 16 weeks, 1 year, 2 years, and 5 years post baseline
  Submaximal cycling test
Muscle strength | Change from baseline to 16 weeks, 1 year, 2 years, and 5 years post baseline
  Upper and lower limb muscle strength
Body mass | Change from baseline to 16 weeks, 1 year, 2 years, and 5 years post baseline
  Scale
Inflammation parameters | Change from baseline to 16 weeks, and 1 year and 5 years post baseline
  Blood
Concentration of Troponin and pro-BNP | Change from baseline to 16 weeks, and 1 year post baseline
  Blood
Muscle cross sectional area | Change from baseline to 16 weeks
  Muscle biopsy
Mitochondrial function, gene activity | Change from baseline to 16 weeks
  Muscle biopsy
Sense of coherence | Baseline
  Sense of coherence questionnaire
Chemotherapy completion | Baseline to 16 weeks
  Relative dose intensity extracted from medical records
Hospitalization | Baseline to 16 weeks
  Hospitalizion rates during chemotherapy extracted from medical records
Blood concentrations | Baseline to 16 weeks
  Neutrophil, lymphocyte, hemoglobin, and platelet concentrations extracted from medical records
Quality adjusted life years | Baseline, 16 weeks, and 1 year post baseline
  Quality adjusted life years based on EORTC-QLQ-C30 (EORTC-8D)
Amsterdam Cognition Scan | 5 years post baseline
  neuropsychological test consisting of 7 computerized online cognitive tests measuring a broad range of cognitive domains, including attention, verbal memory and executive functioning. The score range is between -15 to 50. A higher score indicates a better outcome.
Presence of heart failure | 5 years post baseline
  ECG to assess abnormalities such as left ventricular hypertrophy and/or arrhythmias
Overall survival (OS) | 8 years post baseline
  Register-based overall survival (STEEP Guidelines 2.0): proportion of patients who are still alive at 8 years.
Invasive breast cancer-free survival (IBCFS) | 8 years post baseline
  Register-based invasive breast cancer-free survival (STEEP Guidelines 2.0): proportion of patients who have not developed invasive breast cancer 8 years post-baseline
Breast cancer-specific survival (BCSS) | 8 years post baseline
  Register-based Breast cancer-specific survival (STEEP Guidelines 2.0): the proportion of patients who have survived without dying from breast cancer 8 years post baseline.
Breast cancer-free interval (BCFI) | 8 years post baseline
  Register-based breast cancer-free interval (STEEP Guidelines 2.0): the proportion of patients who have not experienced a breast cancer recurrence 8 years following baseline.
Distant recurrence-free interval (DRFI) | 8 years post baseline
  Register-based distant recurrence-free interval (STEEP Guidelines 2.0): the proportion of patients who have not experienced a distant recurrence within 8 years following baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Wengstrom, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Ansund J, Mijwel S, Bolam KA, Altena R, Wengstrom Y, Rullman E, Rundqvist H. High intensity exercise during breast cancer chemotherapy - effects on long-term myocardial damage and physical capacity - data from the OptiTrain RCT. Cardiooncology. 2021 Feb 15;7(1):7. doi: 10.1186/s40959-021-00091-1. PMID 33588948
- [Derived] Hiensch AE, Mijwel S, Bargiela D, Wengstrom Y, May AM, Rundqvist H. Inflammation Mediates Exercise Effects on Fatigue in Patients with Breast Cancer. Med Sci Sports Exerc. 2021 Mar 1;53(3):496-504. doi: 10.1249/MSS.0000000000002490. PMID 32910094
- [Derived] Bolam KA, Mijwel S, Rundqvist H, Wengstrom Y. Two-year follow-up of the OptiTrain randomised controlled exercise trial. Breast Cancer Res Treat. 2019 Jun;175(3):637-648. doi: 10.1007/s10549-019-05204-0. Epub 2019 Mar 26. PMID 30915663
- [Derived] Mijwel S, Backman M, Bolam KA, Jervaeus A, Sundberg CJ, Margolin S, Browall M, Rundqvist H, Wengstrom Y. Adding high-intensity interval training to conventional training modalities: optimizing health-related outcomes during chemotherapy for breast cancer: the OptiTrain randomized controlled trial. Breast Cancer Res Treat. 2018 Feb;168(1):79-93. doi: 10.1007/s10549-017-4571-3. Epub 2017 Nov 14. PMID 29139007
- [Derived] Wengstrom Y, Bolam KA, Mijwel S, Sundberg CJ, Backman M, Browall M, Norrbom J, Rundqvist H. Optitrain: a randomised controlled exercise trial for women with breast cancer undergoing chemotherapy. BMC Cancer. 2017 Feb 6;17(1):100. doi: 10.1186/s12885-017-3079-x. PMID 28166765